CLINICAL TRIAL: NCT00933959
Title: A Pilot Study of Two Contrasting Intervention Programs for Sleep Management
Brief Title: Pilot Study on Sleep Management for US Veterans
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Gavin West, M.D., SLC VA Medical Center/University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27522
Record Dates: First submitted 2009-06-18; First posted 2009-07-08 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Insomnia
Keywords: Sleep problems; Awareness training program; Mind body bridging
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Parasomnias

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mind-Body Bridging Program (Experimental): Subjects will undergo two approximately 1.5 hr training sessions using MBBP spaced one week apart at the VASLCHCS. Each training session will comprise a number of objectives:
  Session 1:
  1. The patient will discover the underlying cause of the insomnia.
  2. The patient will learn how to use easy to apply tools to quieten the mind to sleep soundly.
  Session 2:
  1. The patient will learn how to reduce daytime stress.
  2. The patient will experience a greater sense of self.
  To be maximally effective, the participant should master these objectives and practice MBBP on a daily basis. Bridging and all the other MBBP techniques can be implemented at any time throughout the day and right up to the onset of sleep.
  Interventions: Behavioral: Mind-Body Bridging Program
- Sleep Hygiene (Active Comparator): Participants in the sleep hygiene arm will receive a 1 hr class directing them to the importance of following a list of up to 15 points (tips) for getting to sleep. These points include: limiting alcohol and caffeine intake before bed, using the bed only for sleeping, and having regular bedtimes. Once the instructor has gone over this list and has described in detail each of the 15 points, the class will have an opportunity to ask questions. The participant will be encouraged to learn and practice the objectives of the sleep hygiene class on a daily basis.
  Interventions: Behavioral: Sleep Hygiene

INTERVENTIONS:
Behavioral: Mind-Body Bridging Program — Bridging aims to reduce the impact of negative thought patterns that contribute to stress in the body.
  Other Names: MBBP
  Arms: Mind-Body Bridging Program
Behavioral: Sleep Hygiene — Treatment as usual
  Other Names: SH
  Arms: Sleep Hygiene

SUMMARY:
The aim of the proposed pilot study is to scientifically evaluate the use of Mind-Body Bridging Program (MBBP) as an effective intervention for improving health outcomes in veterans exhibiting sleep disturbance in the Primary Care Clinic at the Veterans Administration Salt Lake City Health Care System (VASLCHCS).

DETAILED DESCRIPTION:
Participants will be randomly assigned to either MBBP or a treatment as usual sleep hygiene (SH) group. The interventions will last two weeks in which participants will attend 2 classes 1-1.5 hr each over two consecutive weeks. Assessment of the effects of the treatments will be based on self-report outcome measures; participants will complete five questionnaires approximately one week prior to the start of the interventions (pre-treatment) and one week after the second session (post-treatment). The sleep quality assessment questionnaire will be additionally completed after the first session (Week 1).

ELIGIBILITY:
Inclusion Criteria:

1. Selection of subjects will be based on the patients exhibiting sleep disturbance as assessed by a standardized sleep questionnaire. Because we are also interested in the effects of MBBP on co-morbid illnesses besides insomnia, we will include subjects that are being treated for depression, pain, and general medical conditions, except as defined as exclusion criteria. Subjects using anti-depressants, sleep and pain medications, and other medications for any condition that is not under exclusion criteria will be admitted to the study. Thus our inclusion criteria will be broader than those based on DSM-IV for primary insomnia.
2. On the day of the study session, patients must arrive before the session for intervention assignment and to turn in their packets, and thereafter on the same day they must be able to attend a mind-body bridging program or sleep hygiene class (see Study Procedure). In addition, they must also be able to attend the second session the following week.

Exclusion Criteria:

1. The patient presents with significant mental health issues, such as severe psychosis or major depression (as verified by the primary care provider) or the patient is under intensive mental health case management.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Medical Outcomes Study-Sleep Scale | Pre-treatment, Week 1, Post treatment
Medical Outcomes Study Short Form-36 for Veterans | Pre-treatment, Post treatment

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale | Pre-treatment, Post treatment
Five-factor Mindfulness Questionnaire | Pre-treatment, Post treatment
PTSD Check List-Military | Pre-treatment, Post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gavin West, M.D., Principal Investigator — Salt Lake City VA/University of Utah
Locations (1):
- SLC VA Medical Center, Salt Lake City, Utah, United States